CLINICAL TRIAL: NCT00271167
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study to Evaluate Tolerability, Safety, Pharmacokinetics and Efficacy of Intravenous INO-1001 in High Risk Subjects Undergoing Cardiopulmonary Bypass for Coronary Revascularization and/or Valve Surgery.
Brief Title: A Trial of INO-1001 in Patients Undergoing Heart Surgery That Involves Heart-lung Bypass
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: It was determined that the study was not appropriate for demonstrating therapeutic benefit in the cardiopulmonary bypass patient population.
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IPC-05-2004
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Heart Diseases; Postoperative Complications
Keywords: Cardiac surgery; PARP inhibitor; PARP inhibition; Bypass surgery; CPB surgery; Cardiopulmonary bypass; Coronary revascularization; Cardiac valve replacement
MeSH Terms: conditions — Heart Diseases; Postoperative Complications | interventions — INO 1001

INTERVENTIONS:
Drug: INO-1001

SUMMARY:
The purpose of this study is to assess the safety of INO-1001, an intravenous PARP (poly-[ADP ribose] polymerase) inhibitor, in patients undergoing heart surgery. The study also measures whether INO-1001 reduces the side effects caused by heart-lung bypass machines.

DETAILED DESCRIPTION:
Heart-lung bypass during heart surgery sometimes leads to side effects or complications after surgery.

Studies have shown that PARP inhibitors protect cells from damage due to lack of oxygen. Heart-lung bypass during heart surgery can result in cells being deprived of oxygen. INO-1001 may be able to protect these cells and reduce complications following surgery.

A total of 162 patients will be randomly assigned to either INO-1001 or placebo (sugar water). Treatment will begin on the day of heart surgery and continue for 36 hours. A total of 4 doses of INO-1001 will be given. Patients will be followed up until 30 days after surgery.

The following information will be collected: symptoms, vital signs, physical examination, blood and urine tests, electrocardiograms, and other information from medical charts.

The information provided in this listing is disclosed solely to comply with regulatory requirements. The drug INO-1001 has not yet been approved for marketing and is only available to patients who participate in a clinical trial and are chosen for the treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo cardiopulmonary bypass for coronary revascularization and/or valve surgery
* Males and non-pregnant, non-lactating females

Exclusion Criteria:

* Subjects will be required to undergo a full medical review in order to exclude serious medical or psychological illness prior to inclusion
* History of a hypersensitivity reaction to more than three drugs or to mannitol
* Participation in any other investigational study within 30 days of the screening phase
* Known alcohol or drug abuse within the last year
* Treatment with certain restricted medications within a specified time prior to participation in the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162
Dates: Start 2005-10; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Reduction in serious post-operative complications occurring in the first thirty days after surgery.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Methodist Hospital, Houston, Texas
- Australia (4):
  - Sydney, New South Wales
  - Ashford Cardiac Clinic / Adelaide Cardiac, Adelaide, South Australia
  - St. Vincent's Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- India (2):
  - Care Hospital, Hyderabad
  - Escorts Heart Institute and Research Centre, New Delhi
- Israel (2):
  - Wolfson Medical Centre, Holon
  - Jerusalem

REFERENCES:
- [Background] Khan TA, Ruel M, Bianchi C, Voisine P, Komjati K, Szabo C, Sellke FW. Poly(ADP-ribose) polymerase inhibition improves postischemic myocardial function after cardioplegia-cardiopulmonary bypass. J Am Coll Surg. 2003 Aug;197(2):270-7. doi: 10.1016/S1072-7515(03)00538-6. PMID 12892811
- [Background] Virag L, Szabo C. The therapeutic potential of poly(ADP-ribose) polymerase inhibitors. Pharmacol Rev. 2002 Sep;54(3):375-429. doi: 10.1124/pr.54.3.375. PMID 12223530
- [Background] Szabo C. Pharmacological inhibition of poly(ADP-ribose) polymerase in cardiovascular disorders: future directions. Curr Vasc Pharmacol. 2005 Jul;3(3):301-3. doi: 10.2174/1570161054368553. PMID 16026326